## 01/OCT/2016

## Statistical Analysis Plan

Assessment of intercostal block scheduling in preventing acute surgical and post-surgical pain in thoracoscopic surgery

Entrepreneur : Dr. Dan Levy Faber

Address: Medical cente Carmel St. Michel 7, Haifa, 34362

Site of the study: Department Surgery chest House Patients Carmel

Principle Investigator: Dr. Dan Levy Faber

## Statistical analysis

The difference in the number of hospitalization days between the two study populations will be examined in a double-tailed T test. Differences in the proportions of the categorical complications between the two study populations, as well as differences in the pain level, will be examined in the live-squared test as well as in the two-tailed Z proportion test. The significance level is P < 0.05.